CLINICAL TRIAL: NCT01022892
Title: Contrast Ultrasound in the Surveillance of Endovascular Abdominal Aortic Aneurysm Repair
Status: Completed | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Dr. Sudhir Nagpal, Vascular Surgeon, Ottawa Hospital Research Institute
Other Study IDs: 2007607-01H
Record Dates: First submitted 2009-11-26; First posted 2009-12-01 (Estimated); Last update posted 2012-03-07 (Estimated); Status verified 2012-03

CONDITIONS: Endovascular Abdominal Aortic Aneurysm Repair
Keywords: Endovascular; Abdominal; Aortic; Aneurysm; Repair; Surveillance; EVAR; CT; Scan; Endoleaks; Contrast; Enhanced; Ultrasound; Definity; AAA; imaging; No Endoleaks
MeSH Terms: conditions — Aneurysm; Endoleak

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Phase 1 - Pilot phase: Total of 10 patients currently undergoing EVAR Surveillance. These 10 patients include 5 patients with endoleak known from a recent CT scan and 5 patients with no endoleak and shrinking aneurysm.
- Phase 2 - Blinded from CT Scan: This phase of study involves recruitment of 150 patients currently under post-EVAR surveillance. The physicians and ultrasound technologists will be blinded to the result of the CT Scan when performing and interpreting the CUS. The current schedule for EVAR Surveillance will be maintained so that an individual may receive more than one enhanced CT Scan and CUS during the 18 months of the study.

SUMMARY:
The purpose of this study is to support the suspected expectation that Contrast enhanced Ultrasound (CUS) detects all endoleaks that have been detected by Computed Tomography (CT), and also find a number of leaks missed by CT.

The investigators' primary goal is to detect no difference between CT and CUS and provide evidence that CUS is a possible alternative to CT.

ELIGIBILITY:
Inclusion Criteria:

* All patients who underwent EVAR at The Ottawa Hospital and currently under post-EVAR surveillance at The Ottawa Hospital.

Exclusion Criteria:

* Unable to consent for injection of contrast
* Unable to acquire IV access
* Right-to-left, bi-directional, or transient right-to-left cardiac shunts
* Severe pulmonary disease
* Previous hypersensitivity to DEFINITY® or its components
* Unable to be followed as a outpatient by the Vascular Diagnostic Center

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All patients who underwent EVAR at The Ottawa Hospital and are currently undergoing post-EVAR surveillance will be eligible for the study.
Sampling Method: Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2009-09; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sudhir Nagpal, MD, Principal Investigator — The Ottawa Hospital - Division of Vascular & Endovascular Surgery